CLINICAL TRIAL: NCT00283088
Title: Phase 1 Study of Intravenous Thrombolysis Plus Hypothermia for Acute Treatment of Ischemic Stroke
Brief Title: Intravenous Thrombolysis Plus Hypothermia for Acute Treatment of Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Patrick Lyden, MD, Director, UCSD Stroke Center,, University of California San Diego, Stroke Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P50NS44148LYDEN; P50NS044148 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
Keywords: stroke; hypothermia; cooling; tissue plasminogen activator; tPA; thrombolysis
MeSH Terms: conditions — Stroke; Hypothermia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Active Comparator): Groups 1 and 2: Parallel groups, randomized to hypothermia or no hypothermia. Both groups receive tPA as a part of standard of care.
  Interventions: Drug: tissue plasminogen activator
- Group 2 (Active Comparator): Groups 1 and 2: Parallel groups, randomized to hypothermia or no hypothermia. Both groups receive tPA as a part of standard of care.
  Interventions: Procedure: hypothermia; Drug: tissue plasminogen activator
- Group 3 (No Intervention): Groups 3, 4, 5 and 6: Factorial groups, randomized to hypothermia plus tPA, hypothermia alone, tPA alone, or no treatment assignment (standard of care).
- Group 4 (Active Comparator): Groups 3, 4, 5 and 6: Factorial groups, randomized to hypothermia plus tPA, hypothermia alone, tPA alone, or no treatment assignment (standard of care).
  Interventions: Drug: tissue plasminogen activator
- Group 5 (Active Comparator): Groups 3, 4, 5 and 6: Factorial groups, randomized to hypothermia plus tPA, hypothermia alone, tPA alone, or no treatment assignment (standard of care).
  Interventions: Procedure: hypothermia
- Group 6 (Active Comparator): Groups 3, 4, 5 and 6: Factorial groups, randomized to hypothermia plus tPA, hypothermia alone, tPA alone, or no treatment assignment (standard of care).
  Interventions: Procedure: hypothermia; Drug: tissue plasminogen activator

INTERVENTIONS:
Procedure: hypothermia — Hypothermia with or without tPA for stroke. Hypothermia is induced using the Celsius Control™ System.
  Subjects are stratified by time to six groups.
  Arms: Group 2; Group 5; Group 6
Drug: tissue plasminogen activator — tPA is a naturally occurring protein that opens blocked arteries by dissolving blood clots
  Arms: Group 1; Group 2; Group 4; Group 6

SUMMARY:
The purpose of this trial is to evaluate if it is safe to use tissue plasminogen activator (tPA) within 6 hours of stroke onset when combined with hypothermia.

DETAILED DESCRIPTION:
A stroke is usually caused by a blockage in one of the arteries that carries blood to the brain. Research has shown that tissue plasminogen activator (tPA)-a naturally occurring protein that opens blocked arteries by dissolving blood clots-activates the body's ability to dissolve recently formed blood clots and reduces or prevents the brain damage caused by a stroke.

The Food and Drug Administration (FDA) has approved the use of tPA for people having a stroke when taken within 3 hours of stroke onset, but not for those who arrive at the hospital more than 3 hours after stroke onset.

Researchers believe that a lower body temperature (hypothermia) may be beneficial while a stroke is happening because hypothermia may prevent further brain injury, or may make the stroke less damaging. In particular, hypothermia may make it possible to use tPA later than 3 hours after a stroke begins. This study will determine if it is safe to use tPA within 6 hours of the start of a stroke when combined with hypothermia.

Patients will receive a standard stroke evaluation, which includes blood tests, a computed tomography (CT) scan, complete physical and neurological examinations, and an electrocardiogram (EKG) to determine eligibility for the study.

Participants will be randomly assigned to a study group based on when their stroke began. Those who arrive at the hospital less than 3 hours from stroke onset will receive tPA alone or tPA with cooling (hypothermia). Those who arrive at the hospital 3 to 6 hours after stroke onset will be assigned to 1 of 4 groups-receiving either tPA alone, tPA with cooling, cooling alone, or standard medical care. Length of participation (including observation after the patient leaves the hospital) is 90 days.

This study is part of the Specialized Program of Translational Research in Acute Stroke (SPOTRIAS), which allows researchers to enhance and initiate translational research that ultimately will benefit stroke patients by treating more patients in less than 2 hours, and finding ways to treat additional patients later.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* All eligibility criteria for t-PA administration for acute ischemic stroke as outlined by the NINDS tPA Guidelines are met with the exception of time from onset
* Stroke onset within 6 hours prior to planned start of tPA
* Any subtype of ischemic stroke with NIHSS < 7 at the time hypothermia begins

Exclusion Criteria:

* Etiology other than ischemic stroke
* Item 1a on NIHSS>1 at the time of enrollment
* Symptoms resolving or NIHSS < 7 at the time hypothermia begins
* Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis, (cryoglobulinemia, Sickle cell disease, serum cold agglutinins), or vasospastic disorders such as Raynaud's or thromboangiitis obliterans.
* Known co-morbid conditions likely to complicate therapy, e.g., end-stage cardiomyopathy, uncompensated arrhythmia, myopathy, liver disease severe enough to elevate bilirubin, history of pelvic or abdominal mass likely to compress inferior vena cava, IVC filters, dementia severe enough to prevent valid consent, end-stage AIDS, known thyroid deficiency, known renal insufficiency likely to impair meperidine (Demerol®) clearance
* Intracerebral hematoma
* Any intraventricular hemorrhage
* SBP > 185 or < 100; DBP > 110 or < 50 mmHg
* Pregnancy in women of child-bearing potential (must have pregnancy test, urine or blood, prior to therapy).
* Medical conditions likely to interfere with patient assessment
* Known allergy to meperidine (Demerol®)
* Currently taking MAO-I class of medication or used within previous 14 days
* Life expectancy < 3 months
* Not likely to be available for long-term follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2003-10; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence and volume of hemorrhage on CT | 48 hours post onset

SECONDARY OUTCOMES:
Incidence of AE and SAE | 90 days post onset
Mortality in both groups testing whether hypothermia improves mortality after stroke | 90 Day
NIHSS at the end of hypothermia | Hour 23.5 +/- 30 minutes of hypothermia
Modified Rankin and NIHSS | 30 and 90days
CT lesion volume | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lyden, MD, Principal Investigator — University of California San Diego, Stroke Center
Locations (7):
- United States (7):
  - Stanford Medical Center, Palo Alto, California
  - University of California San Diego, Thornton Hospital, San Diego, California
  - Scripps Mercy Hospital, San Diego, California
  - University of California San Diego, Hillcrest Medical Center, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Saint Louis University Medical Center, St Louis, Missouri
  - Herman Memorial Hospital, Houston, Texas

REFERENCES:
- [Background] Lyden PD, Allgren RL, Ng K, Akins P, Meyer B, Al-Sanani F, Lutsep H, Dobak J, Matsubara BS, Zivin J. Intravascular Cooling in the Treatment of Stroke (ICTuS): early clinical experience. J Stroke Cerebrovasc Dis. 2005 May-Jun;14(3):107-14. doi: 10.1016/j.jstrokecerebrovasdis.2005.01.001. PMID 17904009
- [Background] Guluma KZ, Hemmen TM, Olsen SE, Rapp KS, Lyden PD. A trial of therapeutic hypothermia via endovascular approach in awake patients with acute ischemic stroke: methodology. Acad Emerg Med. 2006 Aug;13(8):820-7. doi: 10.1197/j.aem.2006.03.559. Epub 2006 Jun 9. PMID 16766740
- [Background] Hemmen TM, Raman R, Guluma KZ, Meyer BC, Gomes JA, Cruz-Flores S, Wijman CA, Rapp KS, Grotta JC, Lyden PD; ICTuS-L Investigators. Intravenous thrombolysis plus hypothermia for acute treatment of ischemic stroke (ICTuS-L): final results. Stroke. 2010 Oct;41(10):2265-70. doi: 10.1161/STROKEAHA.110.592295. Epub 2010 Aug 19. PMID 20724711
- [Background] Hemmen TM, Lyden PD. Induced hypothermia for acute stroke. Stroke. 2007 Feb;38(2 Suppl):794-9. doi: 10.1161/01.STR.0000247920.15708.fa. PMID 17261741